CLINICAL TRIAL: NCT05766137
Title: Comparison of The Post-Extraction Dimensional Alterations Following Ridge Preservation Using Autogenous Partially and Completely Demineralized Dentin Grafts Versus Autogenous Whole-tooth Graft: A Randomized Controlled Clinical Trial
Brief Title: Comparison of The Post-Extraction Dimensional Alterations Following Ridge Preservation Using Autogenous Partially and Completely Demineralized Dentin Grafts Versus Autogenous Whole-tooth Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Osama Abdelwahab Megahed, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DinaAbdelwahabPerio
Record Dates: First submitted 2023-02-14; First posted 2023-03-13 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Socket Preservation, Alveolar Ridge Deficiency, Alveolar Ridge Preservation

STUDY DESIGN:
Intervention Model Description: Parallel-group with allocation ratio of 1:1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: * Blinding of the operator is not applicable.
  * Participants, outcome assessors and biostatistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ridge preservation by filling the socket with autogenous partially demineralized dentin graft (Experimental): 2% HNO3 partial demineralization for 10 minutes
  Interventions: Procedure: Alveolar ridge preservation
- Ridge preservation by filling the socket with autogenous completely demineralized dentin graft (Experimental): 0.6N HCl for 30 minutes for complete demineralization
  Interventions: Procedure: Alveolar ridge preservation
- Ridge preservation by filling the socket with autogenous whole-tooth graft (AWTG). (Active Comparator): After cleaning the tooth, it will be ground using bone mill and AWTG particles will be prepared by immersing tooth particles in basic ethanol for 10 min for disinfection , then washed twice in saline and dried using sterile gauze.
  Interventions: Procedure: Alveolar ridge preservation

INTERVENTIONS:
Procedure: Alveolar ridge preservation — Socket preservation

SUMMARY:
For alveolar ridge preservation after extraction of a non-restorable maxillary non-molar tooth, will the use of Autogenous partially or completely demineralized dentin grafts result in similar ridge dimensions compared to Autogenous whole-tooth graft?

DETAILED DESCRIPTION:
One inevitable consequence of tooth loss is alveolar ridge resorption, which is progressive, irreversible, chronic, and cumulative. For implant placement, adequate dimensions of the alveolar ride housing are essential for proper implant positioning to provide for both implant stability and esthetics. Various procedures have been developed to limit post-extraction dimensional alterations or to restore normal bone dimensions, among which is ridge preservation. Numerous materials have been introduced and compared, nevertheless the best option is yet to be determined. Autogenous bone remains the gold standard for bone grafting, however one cannot ignore its unavoidable drawbacks, with donor site morbidity and the need for additional surgery having the biggest impact, as well as the limited amount that can be harvested and the unpredictable resorption rate. Several other options have been introduced with the aim of overcoming these disadvantages.

promising results have been reported, and the use of autogenous tooth bone graft (ATBG) is gaining popularity, since this material has a structure that closely resembles bone, especially the dentin which is composed of similar inorganic and organic elements, and also has osteoinductive and osteoconductive capacity.

Some studies using mineralized dentin matrix have shown that the material possesses excellent biocompatibility but is less effective than bone derived products in bone formation. On the other hand, several basic animal studies have shown that completely demineralized dentin matrix to be not only biocompatible, but also osteo-inductive, similar to demineralized bone matrix. The degree of demineralization is critical for optimal dentin regeneration; the partially demineralized dentin matrix is thought to have optimal conditions for dentin regeneration. Partial demineralization results in the elimination of the major part of the mineral phase and immunogenic components while retaining a very low fraction of minerals (5-10 wt%), providing an osteoconductive and osteo-inductive scaffold containing several growth factors.

It is agreed upon that nowadays optimizing protocols of demineralization of dentin grafts is necessary for standardization and further studies are required to determine the most suitable conditions of demineralization and particle sizes of dentin grafts for clinical application in implant dentistry. Additionally, more research is required to investigate whether graft preparation in its simplest form is sufficient or whether enhancing the graft with demineralization will result in any clinical significance.

ELIGIBILITY:
Inclusion Criteria:

* Non-molar maxillary teeth indicated for extraction.
* Extraction sockets having no more than 50% of buccal alveolar bone loss were included.
* Patients at least 18 years or older
* Motivated patients, agree to sign informed consent and complete the follow-up period

Exclusion Criteria:

* Infection at the extraction site
* Smokers
* Patients undergoing or having history of radiotherapy, chemotherapy or bisphosphonate therapy.
* Systemic conditions that may compromise healing or bone metabolism (e.g., uncontrolled diabetes, hyperthyroidism).
* Females that are pregnant or are planning to get pregnant during the study course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge width and height changes | 6 months
  Difference in alveolar ridge width and height linear measurements in millimeters between baseline and final CBCT scans after 6 months

SECONDARY OUTCOMES:
Histological assessment | 6 months
  Visual observation of graft remodeling and new bone formation (descriptive measurement)